CLINICAL TRIAL: NCT01036763
Title: Assessment of COPD Therapy From the Physicians Perspective Using Tiotropium as an Example
Brief Title: Assessment of Chronic Obstructive Pulmonary Disease (COPD) Therapy From the Physicians Perspective Using Tiotropium as an Example
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 205.455
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Documentation of successful therapy with tiotropium (Spiriva Respimat; Spiriva (tiotropium 18 mcg capsules)) in COPD patients requiring long-acting bronchodilators: description of the most important outcome parameters according to the physicians assessment to determine the success of therapy. Such data are not yet available.

Also collection of physicians assessments and patients assessments of efficacy and tolerability of Spiriva Respimat, Spiriva (tiotropium 18 mcg capsules).

DETAILED DESCRIPTION:
Study Design:

observational

ELIGIBILITY:
Inclusion criteria COPD patients requiring long-acting bronchodilators according to approved Summary of Product Characteristics (SPC) and guidelines

Exclusion criteria Patients cannot be recruited if any of the general or specific contraindications listed in the Patient information leaflet or the Summary of Product Characteristics applies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Dates: Start 2010-01; Primary Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (352):
- Germany (352):
  - Boehringer Ingelheim Investigational Site 1, Ahrensburg
  - Boehringer Ingelheim Investigational Site 2, Amberg
  - Boehringer Ingelheim Investigational Site 3, Arnstadt
  - Boehringer Ingelheim Investigational Site 4, Auerbach
  - Boehringer Ingelheim Investigational Site 10, Augsburg
  - Boehringer Ingelheim Investigational Site 5, Augsburg
  - Boehringer Ingelheim Investigational Site 6, Augsburg
  - Boehringer Ingelheim Investigational Site 7, Augsburg
  - Boehringer Ingelheim Investigational Site 8, Augsburg
  - Boehringer Ingelheim Investigational Site 9, Augsburg
  - Boehringer Ingelheim Investigational Site 11, Backnang
  - Boehringer Ingelheim Investigational Site 12, Bad Doberan
  - Boehringer Ingelheim Investigational Site 13, Bad Kissingen
  - Boehringer Ingelheim Investigational Site 15, Bad Kötzting
  - Boehringer Ingelheim Investigational Site 16, Bad Kötzting
  - Boehringer Ingelheim Investigational Site 14, Bad Krozingen
  - Boehringer Ingelheim Investigational Site 17, Bad Lippspringe
  - Boehringer Ingelheim Investigational Site 18, Bad Neuenahr-Ahrweiler
  - Boehringer Ingelheim Investigational Site 19, Bad Neustadt an der Saale
  - Boehringer Ingelheim Investigational Site 20, Bad Reichenhall
  - Boehringer Ingelheim Investigational Site 21, Bad Reichenhall
  - Boehringer Ingelheim Investigational Site 22, Bad Sachsa
  - Boehringer Ingelheim Investigational Site 23, Bad Wörishofen
  - Boehringer Ingelheim Investigational Site 24, Baden-Baden
  - Boehringer Ingelheim Investigational Site 25, Ballenstedt
  - Boehringer Ingelheim Investigational Site 26, Bamberg
  - Boehringer Ingelheim Investigational Site 27, Bautzen
  - Boehringer Ingelheim Investigational Site 28, Beelitz
  - Boehringer Ingelheim Investigational Site 29, Bensheim
  - Boehringer Ingelheim Investigational Site 30, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site 31, Berlin
  - Boehringer Ingelheim Investigational Site 32, Berlin
  - Boehringer Ingelheim Investigational Site 33, Berlin
  - Boehringer Ingelheim Investigational Site 34, Berlin
  - Boehringer Ingelheim Investigational Site 35, Berlin
  - Boehringer Ingelheim Investigational Site 36, Berlin
  - Boehringer Ingelheim Investigational Site 37, Berlin
  - Boehringer Ingelheim Investigational Site 38, Berlin
  - Boehringer Ingelheim Investigational Site 39, Berlin
  - Boehringer Ingelheim Investigational Site 40, Berlin
  - Boehringer Ingelheim Investigational Site 41, Berlin
  - Boehringer Ingelheim Investigational Site 42, Berlin
  - Boehringer Ingelheim Investigational Site 43, Berlin
  - Boehringer Ingelheim Investigational Site 44, Berlin
  - Boehringer Ingelheim Investigational Site 45, Berlin
  - Boehringer Ingelheim Investigational Site 46, Berlin
  - Boehringer Ingelheim Investigational Site 47, Berlin
  - Boehringer Ingelheim Investigational Site 48, Berlin
  - Boehringer Ingelheim Investigational Site 49, Berlin
  - Boehringer Ingelheim Investigational Site 50, Berlin
  - Boehringer Ingelheim Investigational Site 51, Berlin
  - Boehringer Ingelheim Investigational Site 52, Berlin
  - Boehringer Ingelheim Investigational Site 53, Bernau
  - Boehringer Ingelheim Investigational Site 54, Bitterfeld-Wolfen
  - Boehringer Ingelheim Investigational Site 55, Bochum
  - Boehringer Ingelheim Investigational Site 56, Bochum
  - Boehringer Ingelheim Investigational Site 57, Bonn
  - Boehringer Ingelheim Investigational Site 58, Bonn
  - Boehringer Ingelheim Investigational Site 59, Bonn
  - Boehringer Ingelheim Investigational Site 60, Bonn
  - Boehringer Ingelheim Investigational Site 61, Bottrop
  - Boehringer Ingelheim Investigational Site 62, Braunschweig
  - Boehringer Ingelheim Investigational Site 63, Braunschweig
  - Boehringer Ingelheim Investigational Site 64, Bremen
  - Boehringer Ingelheim Investigational Site 65, Bremen
  - Boehringer Ingelheim Investigational Site 66, Bremen
  - Boehringer Ingelheim Investigational Site 67, Bremen
  - Boehringer Ingelheim Investigational Site 68, Bremerhaven
  - Boehringer Ingelheim Investigational Site 69, Bremerhaven
  - Boehringer Ingelheim Investigational Site 70, Bruchsal
  - Boehringer Ingelheim Investigational Site 71, Buchholz
  - Boehringer Ingelheim Investigational Site 72, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 73, Celle
  - Boehringer Ingelheim Investigational Site 74, Celle
  - Boehringer Ingelheim Investigational Site 75, Chemnitz
  - Boehringer Ingelheim Investigational Site 76, Coburg
  - Boehringer Ingelheim Investigational Site 77, Coburg
  - Boehringer Ingelheim Investigational Site 200, Cologne
  - Boehringer Ingelheim Investigational Site 201, Cologne
  - Boehringer Ingelheim Investigational Site 202, Cologne
  - Boehringer Ingelheim Investigational Site 78, Cottbus
  - Boehringer Ingelheim Investigational Site 79, Cottbus
  - Boehringer Ingelheim Investigational Site 80, Dachau
  - Boehringer Ingelheim Investigational Site 81, Darmstadt
  - Boehringer Ingelheim Investigational Site 82, Deggendorf
  - Boehringer Ingelheim Investigational Site 83, Delitzsch
  - Boehringer Ingelheim Investigational Site 84, Dessau
  - Boehringer Ingelheim Investigational Site 85, Dillingen
  - Boehringer Ingelheim Investigational Site 86, Dillingen
  - Boehringer Ingelheim Investigational Site 87, Donaueschingen
  - Boehringer Ingelheim Investigational Site 88, Dorsten
  - Boehringer Ingelheim Investigational Site 89, Dortmund
  - Boehringer Ingelheim Investigational Site 90, Dresden
  - Boehringer Ingelheim Investigational Site 91, Dresden
  - Boehringer Ingelheim Investigational Site 92, Dresden
  - Boehringer Ingelheim Investigational Site 93, Dresden
  - Boehringer Ingelheim Investigational Site 94, Dresden
  - Boehringer Ingelheim Investigational Site 95, Dresden
  - Boehringer Ingelheim Investigational Site 96, Dresden
  - Boehringer Ingelheim Investigational Site 97, Düren
  - Boehringer Ingelheim Investigational Site 98, Düren
  - Boehringer Ingelheim Investigational Site 100, Düsseldorf
  - Boehringer Ingelheim Investigational Site 101, Düsseldorf
  - Boehringer Ingelheim Investigational Site 102, Düsseldorf
  - Boehringer Ingelheim Investigational Site 99, Düsseldorf
  - Boehringer Ingelheim Investigational Site 103, Eichstätt
  - Boehringer Ingelheim Investigational Site 104, Emden
  - Boehringer Ingelheim Investigational Site 105, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site 106, Erfurt
  - Boehringer Ingelheim Investigational Site 107, Erfurt
  - Boehringer Ingelheim Investigational Site 108, Erfurt
  - Boehringer Ingelheim Investigational Site 109, Erlangen
  - Boehringer Ingelheim Investigational Site 110, Eschwege
  - Boehringer Ingelheim Investigational Site 111, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site 112, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site 113, Euskirchen
  - Boehringer Ingelheim Investigational Site 114, Fellbach
  - Boehringer Ingelheim Investigational Site 115, Flensburg
  - Boehringer Ingelheim Investigational Site 116, Forchheim
  - Boehringer Ingelheim Investigational Site 123, Föhren
  - Boehringer Ingelheim Investigational Site 117, Frankenthal
  - Boehringer Ingelheim Investigational Site 118, Frankfurt
  - Boehringer Ingelheim Investigational Site 119, Frankfurt
  - Boehringer Ingelheim Investigational Site 120, Frankfurt
  - Boehringer Ingelheim Investigational Site 121, Frankfurt
  - Boehringer Ingelheim Investigational Site 122, Freising
  - Boehringer Ingelheim Investigational Site 124, Fürstenfeldbruck
  - Boehringer Ingelheim Investigational Site 125, Fürth
  - Boehringer Ingelheim Investigational Site 126, Fürth
  - Boehringer Ingelheim Investigational Site 127, Ganderkesee
  - Boehringer Ingelheim Investigational Site 128, Gauting
  - Boehringer Ingelheim Investigational Site 129, Geilenkirchen
  - Boehringer Ingelheim Investigational Site 130, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 131, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 132, Gera
  - Boehringer Ingelheim Investigational Site 133, Germering
  - Boehringer Ingelheim Investigational Site 134, Giessen
  - Boehringer Ingelheim Investigational Site 135, Giessen
  - Boehringer Ingelheim Investigational Site 140, Göppingen
  - Boehringer Ingelheim Investigational Site 141, Göttingen
  - Boehringer Ingelheim Investigational Site 142, Göttingen
  - Boehringer Ingelheim Investigational Site 143, Göttingen
  - Boehringer Ingelheim Investigational Site 136, Greiz
  - Boehringer Ingelheim Investigational Site 137, Grevesmühlen
  - Boehringer Ingelheim Investigational Site 138, Großenhain
  - Boehringer Ingelheim Investigational Site 139, Gummersbach
  - Boehringer Ingelheim Investigational Site 144, Günzburg
  - Boehringer Ingelheim Investigational Site 145, Gütersloh
  - Boehringer Ingelheim Investigational Site 146, Gütersloh
  - Boehringer Ingelheim Investigational Site 147, Gütersloh
  - Boehringer Ingelheim Investigational Site 148, Hagen
  - Boehringer Ingelheim Investigational Site 149, Halberstadt
  - Boehringer Ingelheim Investigational Site 150, Halle
  - Boehringer Ingelheim Investigational Site 151, Halle
  - Boehringer Ingelheim Investigational Site 152, Hamburg
  - Boehringer Ingelheim Investigational Site 153, Hamburg
  - Boehringer Ingelheim Investigational Site 154, Hamburg
  - Boehringer Ingelheim Investigational Site 155, Hamburg
  - Boehringer Ingelheim Investigational Site 156, Hamburg
  - Boehringer Ingelheim Investigational Site 157, Hamburg
  - Boehringer Ingelheim Investigational Site 158, Hamburg
  - Boehringer Ingelheim Investigational Site 159, Hamburg
  - Boehringer Ingelheim Investigational Site 160, Hamburg
  - Boehringer Ingelheim Investigational Site 161, Hamburg
  - Boehringer Ingelheim Investigational Site 162, Hamburg
  - Boehringer Ingelheim Investigational Site 163, Hamm
  - Boehringer Ingelheim Investigational Site 164, Hanover
  - Boehringer Ingelheim Investigational Site 165, Hanover
  - Boehringer Ingelheim Investigational Site 166, Hanover
  - Boehringer Ingelheim Investigational Site 167, Hanover
  - Boehringer Ingelheim Investigational Site 168, Hartha
  - Boehringer Ingelheim Investigational Site 169, Heidelberg
  - Boehringer Ingelheim Investigational Site 170, Heidelberg
  - Boehringer Ingelheim Investigational Site 171, Heidelberg
  - Boehringer Ingelheim Investigational Site 172, Heidelberg
  - Boehringer Ingelheim Investigational Site 173, Heilbronn
  - Boehringer Ingelheim Investigational Site 174, Heilbronn
  - Boehringer Ingelheim Investigational Site 175, Hemmingen
  - Boehringer Ingelheim Investigational Site 176, Hemmingen
  - Boehringer Ingelheim Investigational Site 177, Herne
  - Boehringer Ingelheim Investigational Site 178, Hettstedt
  - Boehringer Ingelheim Investigational Site 179, Hilden
  - Boehringer Ingelheim Investigational Site 180, Husum
  - Boehringer Ingelheim Investigational Site 181, Itzehoe
  - Boehringer Ingelheim Investigational Site 182, Itzehoe
  - Boehringer Ingelheim Investigational Site 183, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 184, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 185, Kamen
  - Boehringer Ingelheim Investigational Site 186, Karlsruhe
  - Boehringer Ingelheim Investigational Site 187, Karlsruhe
  - Boehringer Ingelheim Investigational Site 188, Kempten
  - Boehringer Ingelheim Investigational Site 189, Kiel
  - Boehringer Ingelheim Investigational Site 190, Kiel
  - Boehringer Ingelheim Investigational Site 191, Kiel
  - Boehringer Ingelheim Investigational Site 192, Kirchheim
  - Boehringer Ingelheim Investigational Site 193, Koblenz
  - Boehringer Ingelheim Investigational Site 194, Koblenz
  - Boehringer Ingelheim Investigational Site 195, Koblenz
  - Boehringer Ingelheim Investigational Site 196, Koblenz
  - Boehringer Ingelheim Investigational Site 197, Konstanz
  - Boehringer Ingelheim Investigational Site 203, Königs Wusterhausen
  - Boehringer Ingelheim Investigational Site 204, Köthen
  - Boehringer Ingelheim Investigational Site 198, Krefeld
  - Boehringer Ingelheim Investigational Site 199, Krefeld
  - Boehringer Ingelheim Investigational Site 205, Landshut
  - Boehringer Ingelheim Investigational Site 206, Langen
  - Boehringer Ingelheim Investigational Site 207, Langenfeld
  - Boehringer Ingelheim Investigational Site 208, Langenfeld
  - Boehringer Ingelheim Investigational Site 209, Leipzig
  - Boehringer Ingelheim Investigational Site 210, Leipzig
  - Boehringer Ingelheim Investigational Site 211, Leipzig
  - Boehringer Ingelheim Investigational Site 212, Leonberg
  - Boehringer Ingelheim Investigational Site 213, Leverkusen
  - Boehringer Ingelheim Investigational Site 214, Leverkusen
  - Boehringer Ingelheim Investigational Site 215, Lichtenfels
  - Boehringer Ingelheim Investigational Site 216, Limburg
  - Boehringer Ingelheim Investigational Site 217, Lippstadt
  - Boehringer Ingelheim Investigational Site 221, Loerrach
  - Boehringer Ingelheim Investigational Site 218, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 219, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 222, Lüneburg
  - Boehringer Ingelheim Investigational Site 223, Lüneburg
  - Boehringer Ingelheim Investigational Site 224, Lützen
  - Boehringer Ingelheim Investigational Site 225, Magdeburg
  - Boehringer Ingelheim Investigational Site 226, Magdeburg
  - Boehringer Ingelheim Investigational Site 227, Mainz
  - Boehringer Ingelheim Investigational Site 228, Mainz
  - Boehringer Ingelheim Investigational Site 229, Mannheim
  - Boehringer Ingelheim Investigational Site 230, Mannheim
  - Boehringer Ingelheim Investigational Site 231, Marburg
  - Boehringer Ingelheim Investigational Site 232, Markkleeberg
  - Boehringer Ingelheim Investigational Site 233, Marktredwitz
  - Boehringer Ingelheim Investigational Site 234, Menden
  - Boehringer Ingelheim Investigational Site 235, Minden
  - Boehringer Ingelheim Investigational Site 236, Minden
  - Boehringer Ingelheim Investigational Site 237, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 238, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 239, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 240, Mühlhausen
  - Boehringer Ingelheim Investigational Site 241, München
  - Boehringer Ingelheim Investigational Site 242, München
  - Boehringer Ingelheim Investigational Site 243, München
  - Boehringer Ingelheim Investigational Site 244, München
  - Boehringer Ingelheim Investigational Site 245, München
  - Boehringer Ingelheim Investigational Site 246, München
  - Boehringer Ingelheim Investigational Site 247, München
  - Boehringer Ingelheim Investigational Site 248, München
  - Boehringer Ingelheim Investigational Site 249, Münster
  - Boehringer Ingelheim Investigational Site 250, Münster
  - Boehringer Ingelheim Investigational Site 251, Münster
  - Boehringer Ingelheim Investigational Site 252, Neu-Ulm
  - Boehringer Ingelheim Investigational Site 253, Neumarkt
  - Boehringer Ingelheim Investigational Site 254, Neuwied
  - Boehringer Ingelheim Investigational Site 255, Niesky
  - Boehringer Ingelheim Investigational Site 256, Norderstedt
  - Boehringer Ingelheim Investigational Site 257, Norderstedt
  - Boehringer Ingelheim Investigational Site 258, Nordhausen
  - Boehringer Ingelheim Investigational Site 259, Nuremberg
  - Boehringer Ingelheim Investigational Site 260, Nuremberg
  - Boehringer Ingelheim Investigational Site 261, Nuremberg
  - Boehringer Ingelheim Investigational Site 262, Nuremberg
  - Boehringer Ingelheim Investigational Site 263, Oberursel
  - Boehringer Ingelheim Investigational Site 264, Offenburg
  - Boehringer Ingelheim Investigational Site 265, Olpe
  - Boehringer Ingelheim Investigational Site 266, Oranienburg
  - Boehringer Ingelheim Investigational Site 267, Oschatz
  - Boehringer Ingelheim Investigational Site 268, Oschersleben
  - Boehringer Ingelheim Investigational Site 269, Osnabrück
  - Boehringer Ingelheim Investigational Site 270, Parsberg
  - Boehringer Ingelheim Investigational Site 271, Peine
  - Boehringer Ingelheim Investigational Site 272, Pforzheim
  - Boehringer Ingelheim Investigational Site 273, Plauen
  - Boehringer Ingelheim Investigational Site 274, Plauen
  - Boehringer Ingelheim Investigational Site 275, Plauen
  - Boehringer Ingelheim Investigational Site 276, Potsdam
  - Boehringer Ingelheim Investigational Site 277, Pulheim
  - Boehringer Ingelheim Investigational Site 278, Rathenow
  - Boehringer Ingelheim Investigational Site 279, Ratingen
  - Boehringer Ingelheim Investigational Site 280, Raubach
  - Boehringer Ingelheim Investigational Site 281, Regensburg
  - Boehringer Ingelheim Investigational Site 282, Remscheid
  - Boehringer Ingelheim Investigational Site 283, Remscheid
  - Boehringer Ingelheim Investigational Site 284, Rostock
  - Boehringer Ingelheim Investigational Site 285, Rostock
  - Boehringer Ingelheim Investigational Site 286, Roth
  - Boehringer Ingelheim Investigational Site 287, Rottach-Egern
  - Boehringer Ingelheim Investigational Site 288, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site 289, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site 290, Saalfeld
  - Boehringer Ingelheim Investigational Site 291, Saarbrücken
  - Boehringer Ingelheim Investigational Site 292, Saarbrücken
  - Boehringer Ingelheim Investigational Site 293, Saarbrücken
  - Boehringer Ingelheim Investigational Site 294, Saarbrücken
  - Boehringer Ingelheim Investigational Site 295, Saarbrücken
  - Boehringer Ingelheim Investigational Site 296, Saarlouis
  - Boehringer Ingelheim Investigational Site 297, Saarlouis
  - Boehringer Ingelheim Investigational Site 314, Saint Ingbert
  - Boehringer Ingelheim Investigational Site 298, Salzgitter
  - Boehringer Ingelheim Investigational Site 299, Schmallenberg
  - Boehringer Ingelheim Investigational Site 300, Schmölln
  - Boehringer Ingelheim Investigational Site 301, Schmölln
  - Boehringer Ingelheim Investigational Site 302, Schwabach
  - Boehringer Ingelheim Investigational Site 303, Schwandorf in Bayern
  - Boehringer Ingelheim Investigational Site 305, Schwäbisch Gmünd
  - Boehringer Ingelheim Investigational Site 304, Schwedt
  - Boehringer Ingelheim Investigational Site 306, Sebnitz
  - Boehringer Ingelheim Investigational Site 307, Seevetal
  - Boehringer Ingelheim Investigational Site 308, Siegen
  - Boehringer Ingelheim Investigational Site 309, Simmern
  - Boehringer Ingelheim Investigational Site 310, Sinsheim
  - Boehringer Ingelheim Investigational Site 311, Solingen
  - Boehringer Ingelheim Investigational Site 312, Sondershausen
  - Boehringer Ingelheim Investigational Site 313, Sonneberg
  - Boehringer Ingelheim Investigational Site 315, Stade
  - Boehringer Ingelheim Investigational Site 316, Stadthagen
  - Boehringer Ingelheim Investigational Site 317, Starnberg
  - Boehringer Ingelheim Investigational Site 318, Starnberg
  - Boehringer Ingelheim Investigational Site 319, Staufen
  - Boehringer Ingelheim Investigational Site 320, Steinbach
  - Boehringer Ingelheim Investigational Site 321, Steinhagen
  - Boehringer Ingelheim Investigational Site 322, Steinhagen
  - Boehringer Ingelheim Investigational Site 323, Strausberg
  - Boehringer Ingelheim Investigational Site 324, Straußfurt
  - Boehringer Ingelheim Investigational Site 325, Stuttgart
  - Boehringer Ingelheim Investigational Site 326, Stuttgart
  - Boehringer Ingelheim Investigational Site 327, Stuttgart
  - Boehringer Ingelheim Investigational Site 328, Stuttgart
  - Boehringer Ingelheim Investigational Site 329, Teltow
  - Boehringer Ingelheim Investigational Site 330, Teterow
  - Boehringer Ingelheim Investigational Site 331, Teuchern
  - Boehringer Ingelheim Investigational Site 332, Troisdorf
  - Boehringer Ingelheim Investigational Site 333, Ulm
  - Boehringer Ingelheim Investigational Site 334, Uttenreuth
  - Boehringer Ingelheim Investigational Site 335, Waiblingen
  - Boehringer Ingelheim Investigational Site 336, Waren
  - Boehringer Ingelheim Investigational Site 337, Weilheim
  - Boehringer Ingelheim Investigational Site 338, Weyhe
  - Boehringer Ingelheim Investigational Site 339, Wiesbaden
  - Boehringer Ingelheim Investigational Site 340, Wiesbaden
  - Boehringer Ingelheim Investigational Site 341, Wiesloch
  - Boehringer Ingelheim Investigational Site 342, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 343, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 344, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 345, Witten
  - Boehringer Ingelheim Investigational Site 346, Witten
  - Boehringer Ingelheim Investigational Site 347, Witten
  - Boehringer Ingelheim Investigational Site 220, Wittenberg
  - Boehringer Ingelheim Investigational Site 348, Wolfsburg
  - Boehringer Ingelheim Investigational Site 349, Wolfsburg
  - Boehringer Ingelheim Investigational Site 350, Würzburg
  - Boehringer Ingelheim Investigational Site 351, Zerbst
  - Boehringer Ingelheim Investigational Site 352, Zirndorf

REFERENCES:
- [Background] Rau-Berger H, Kroker A, Mitfessel H, Schmidt H, Glaab T Assessment of COPD-therapy with tiotropium by the treating pneumologist. 53rd Cong of the German Respiratory Society, Nuremberg, 29 Mar - 1 Apr 2012 (Poster), (2012)
- [Background] Glaab T, Kroker A, Mitfessel H, Schmdit H, Rau-Berger H Evaluation of COPD treatment success by office-based pneumologists using the example of tiotropium. 21st Ann Cong of the European Respiratory Society (ERS), Amsterdam, 24 - 28 Sep 2011 (Poster), (2011)

RESULTS

PARTICIPANT FLOW:
Groups:
- Spiriva® 18 Microgram/Spiriva® Respimat®: 1 capsule/2 puffs once daily at the same time
Period: Overall Study
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Started | 1264
Completed | 1171
Not Completed | 93
Not completed — Adverse Event | 25
Not completed — Lost to Follow-up | 28
Not completed — Other reason (not specified) | 40

BASELINE CHARACTERISTICS:
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Number analyzed (Participants) | 1264
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (10.5)
Age, Customized [Number; unit: Years]
  < 65 years | 569
  >= 65 years | 695
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 466
  Male | 798

OUTCOME MEASURES:

1. Primary Outcome: Success of Treatment With Tiotropium According to Physician's Assessment
Description: Evaluation of important outcome parameters (pulmonary function, dyspnoe, health-related quality of life, exercise capacity, prevention of exacerbations) which were used for the physician´s decision to assess the treatment as successful
Time Frame: 6 - 12 weeks
Population: All patients who were documented to have taken at least one dose of Spiriva®18 Microgram/Spiriva® Respimat® and had COPD requiring long-acting anticholinergics
Measure: Number; unit: Participants
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Number analyzed (Participants) | 1264
Participants
  Pulmonary function | 620
  Exercise capacity | 618
  Dyspnoea | 452
  Quality of life | 412
  Patient's opinion | 235
  Prevention of exacerbations | 106

2. Primary Outcome: Assessment of Efficacy According to Physician
Description: Physician's assessment of efficacy within categories (positive/ negative), concurrent proportion of positive efficacy assessments by both physician and patient was determined
Time Frame: 6 - 12 weeks
Measure: Number; unit: Participants
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Number analyzed (Participants) | 1264
Participants
  Very good | 342
  Good | 645
  Satisfactory | 172
  Less satisfactory | 44
  Unsatisfactory | 27
  Missing | 34

3. Primary Outcome: Assessment of Tolerability According to Physician
Description: Physician's assessment of tolerability (positve/ negative), concurrent proportion of positive efficacy assessments by both physician and patient was determined
Time Frame: 6 - 12 weeks
Measure: Number; unit: Participants
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Number analyzed (Participants) | 1264
Participants
  Very good | 601
  Good | 572
  Satisfactory | 35
  Less satisfactory | 9
  Unsatisfactory | 13
  Missing | 34

4. Primary Outcome: Assessment of Efficacy According to Patient
Description: patient-reported assessment within categories (Very good, good, satisfactory, less satisfactory, unsatisfactory, missing)
Time Frame: 6 - 12 weeks
Measure: Number; unit: Participants
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Number analyzed (Participants) | 1264
Participants
  Very good | 339
  Good | 620
  Satisfactory | 169
  Less satisfactory | 55
  Unsatisfactory | 35
  Missing | 46

5. Primary Outcome: Assessment of Tolerability According to Patient
Description: as for outcome 4
Time Frame: 6 - 12 weeks
Measure: Number; unit: Participants
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Number analyzed (Participants) | 1264
Participants
  Very good | 564
  Good | 567
  Satisfactory | 54
  Less satisfactory | 14
  Unsatisfactory | 17
  Missing | 48

6. Secondary Outcome: Physician's Global Evaluation at Visit 1
Description: Physician's global evaluation (PGE) of the patients' general condition at Visit 1 evaluated on an 8-point scale with the scores "Poor (1, 2)", "Satisfactory (3, 4)", "Good (5, 6)" and "Excellent (7, 8)" prior to treatment with Spiriva.
Time Frame: 0 weeks
Measure: Number; unit: Participants
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Number analyzed (Participants) | 1264
Participants
  Excellent | 8
  Good | 294
  Satisfactory | 755
  Poor | 206
  Missing | 1

7. Secondary Outcome: Physician's Global Evaluation at Visit 2
Description: Physician's global evaluation (PGE) of the patients' general condition at Visit 2 evaluated on an 8-point scale after approximately 6-12 weeks of treatment with Spiriva.
Time Frame: after 6 - 12 weeks
Measure: Number; unit: Participants
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Number analyzed (Participants) | 1264
Participants
  Excellent | 61
  Good | 737
  Satisfactory | 407
  Poor | 31
  Missing | 28

ADVERSE EVENTS:
Time Frame: 6 - 12 weeks
Arm/Group | Spiriva® 18 Microgram/Spiriva® Respimat®
Serious Adverse Events (participants affected / at risk) | 5/1264
Other Adverse Events (participants affected / at risk) | 0/1264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva® 18 Microgram/Spiriva® Respimat® (N=1264)
Coronary artery disease (Cardiac disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Condition aggravated (General disorders) | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.